CLINICAL TRIAL: NCT07276113
Title: Enriched Eggs as a Sustainable Approach to Enhance Omega-3 Status in Elite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Matthew Hooks, Mr, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MHLS 23_68
Record Dates: First submitted 2025-11-20; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Suboptimal Omega-3 Index

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): omega-3 enriched egg (14 eggs weekly for 8 weeks, ~250mg DHA daily).
  Interventions: Other: omega-3 enriched eggs
- Control (Placebo Comparator): Non enriched egg group (14 eggs per week for 8 weeks)
  Interventions: Other: non-enriched eggs

INTERVENTIONS:
Other: omega-3 enriched eggs — omega-3 enriched eggs
  Arms: Intervention
Other: non-enriched eggs — non-omega-3 enriched eggs
  Arms: Control

SUMMARY:
The study looked to identify the benefit of omega-3 enriched eggs on circulating omega-3 fatty acid profile of elite level athletes

DETAILED DESCRIPTION:
Study hypothesis: Consuming omega-3 enriched eggs (compared to control) will (1) increase omega-3 index whilst also (2) improving subjective markers of recovery and other health parameters.

Aims & objective:

Overall aim: To investigate the impact of consuming omega-3 enriched eggs blood fatty acid profile among elite level athletes who do not reach omega-3 index targets of 8%, compared to control. Secondary data collected will analyse the impact on health and recovery parameters.

Primary objective: To assess the effect of consuming omega-3 enriched eggs on blood fatty acid response (omega-3 index) in elite level athletes.

Secondary objective: To assess the effect of consuming omega-3 enriched eggs on subjective recovery markers using validated questionnaires (RESTQ-Sport-36, appendix 1; Acute Recovery & Stress Scale, appendix 2) and other health parameters including resting heart rate and blood pressure.

Recruitment Participants will be recruited from Sport Ireland Institute of Sport (SII). SII are partners for this PhD and will provide access for recruitment to those teams/ athletes based in Dublin. Further recruitment will be open to teams across the island of Ireland where potential participants are competing at the highest level within that sport. All relevant permissions will be obtained before commencing any recruitment strategy. All recruitment will initially require approval from the Head of Performance for that sport, this will allow for the researcher to provide athletes with an information sheet, screening questionnaire and consent form. Secondary recruitment will be via a poster which will be put up around the campus. This recruitment will be provided approval by relevant individuals in SII and QUB. The poster will have a QR code which links the interested party to the participant information sheet and screening questionnaire.

Primary objective data collection:

Participants from both omega-3 enriched group and control group will provide a dried blood spot at week 0 (before starting intervention) and post 8-week intervention. The first step is to increase blood flow to the hands; this is done by asking the participant to wash their hands in warm water. The tip of the index finger is prepared with an antibacterial wipe, and this is allowed to dry unassisted. A lancet is then used to draw blood with the first show of blood being wiped away with gauze. The finger is gently squeezed, allowing a blood drop to form. The blood drop is allowed to drop onto the designated spot of the collection card. The collection cards are pre-treated with a proprietary antioxidant treatment called OxyStop, this prevents oxidative loss of PUFAs. The sample is allowed to dry for a few minutes before being sent the same day to a commercial laboratory for analysis (OmegaQuant, University of Stirling, GB).

Co-investigators are familiar with collecting OmegaQuant blood samples through previous professional experience.

ELIGIBILITY:
Inclusion Criteria:

• Participants must be elite level female athletes (tier 4 or 5)

Exclusion Criteria:

* Non-smokers
* Must not be taking statins to lower LDL cholesterol levels.
* Must not have high blood pressure (systolic >140/ diastolic >90mmHg)
* Participants must remain injury free (not miss training >1week)
* Baseline omega-3 index of <8%
* Currently include eggs as part of their habitual diet.
* Participants must be willing to consume 14 eggs per week for 8 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
omega-3 index | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nugent, Doctorate, Principal Investigator — Queens University Belfast
Locations (2):
- Sport Ireland Institute, Dublin, Dublin, Ireland
- Garvaghey Centre, Omagh, Tyrone, United Kingdom

IPD SHARING:
Plan to Share IPD: No